CLINICAL TRIAL: NCT00045474
Title: Phase I Brachytherapy Dose Escalating Study Using the Proxima Therapeutics, Inc. GliaSite RTS in Patients With Recurrent Malignant Gliomas
Brief Title: Brachytherapy in Treating Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000256587; NABTT-2106; JHOC-NABTT-2106
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2003-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult glioblastoma; recurrent adult brain tumor; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Oligodendroglioma; Glioblastoma; Brain Neoplasms; Gliosarcoma | interventions — Chemotherapy, Adjuvant; Iodine-125

INTERVENTIONS:
Procedure: adjuvant therapy
Radiation: iodine I 125

SUMMARY:
RATIONALE: Brachytherapy uses radioactive material to kill cancer cells remaining after surgery.

PURPOSE: Phase I trial to study the effectiveness of brachytherapy in treating patients who have recurrent malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of brachytherapy using an intracavitary applicator and liquid iodine I 125 in patients with recurrent malignant glioma.
* Determine the acute and chronic toxicity of this therapy in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Within 3-21 days after surgical resection, patients receive brachytherapy using an intracavity balloon application (GliaSite) with iodine I 125 solution for a total of 5-7 days.

Cohorts of 5-10 patients receive escalating doses of brachytherapy until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 10 patients experience dose-limiting toxicity.

Patients are followed at 4 weeks and then every 2 months for 1 year.

PROJECTED ACCRUAL: Approximately 20-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant glioma

  * Anaplastic astrocytoma, anaplastic oligodendroglioma, or glioblastoma multiforme

    * Low-grade astrocytoma that progresses to high-grade astrocytoma allowed
  * Unifocal disease
  * Progressive or recurrent after radiotherapy with or without chemotherapy

    * Previously treated with at least 5,000 cGy external beam radiotherapy more than 3 months ago
* Candidate for maximal surgical resection

  * Any expected residual enhancing tumor must be within expected brachytherapy treatment volume
  * Resection must not be expected to result in a new permanent neurologic deficit
* No tumor crossing more than 1 cm beyond the midline on preoperative MRI or CT scan
* No grossly or radiographically apparent leptomeningeal spread
* No ventricular invasion outside the anticipated radiotherapy treatment volume
* No marked edema on MRI or CT scan
* Patients with 2 or more separate foci of contrast-enhancing tumors that are more than 5 cm apart on preoperative MRI or CT scan are ineligible

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Not specified

Renal

* Creatinine no greater than 1.7 mg/dL
* BUN no greater than 2 times upper limit of normal

Cardiovascular

* No uncontrolled hypertension
* No unstable angina pectoris
* No uncontrolled cardiac dysrhythmia

Other

* Mini mental score at least 15
* No other medical illness that would preclude study participation
* No serious infection
* No other malignancy within the past 5 years except curatively treated carcinoma in situ of the cervix or nonmelanoma skin cancer
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy
* No concurrent biologic agents (e.g., immunotoxins, immunoconjugates, antiangiogenesis compounds, antisense therapy, peptide receptor antagonists, interferons, interleukins, tumor-infiltrating lymphocytes, lymphokine-activated killer cells, or gene therapy)

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No concurrent polifeprosan 20 with carmustine implant (Gliadel wafer)

Endocrine therapy

* Concurrent corticosteroids allowed to improve quality of life

Radiotherapy

* See Disease Characteristics
* No concurrent radiosurgery

Surgery

* See Disease Characteristics
* See Radiotherapy

Other

* Recovered from prior therapy
* No prior investigational agents
* No investigational agents during and for 90 days after study participation
* Concurrent cytotoxic treatment allowed to improve quality of life

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10

CONTACTS AND LOCATIONS:
Overall Officials: Larry Kleinberg, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (9):
- United States (9):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abramson Cancer Center at University of Pennsylvania Medical Center, Philadelphia, Pennsylvania